CLINICAL TRIAL: NCT02761382
Title: Mindfulness-based Psychological Pain Treatment in Endometriosis
Brief Title: Psychological Pain Treatment in Endometriosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); TrygFonden, Denmark (Industry); Copenhagen University Hospital, Denmark (Other); Endometriose Foreningen (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AUENDO
Record Dates: First submitted 2016-04-12; First posted 2016-05-04 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2018-06

CONDITIONS: Endometriosis; Pelvic Pain; Chronic Pain
MeSH Terms: conditions — Endometriosis; Pelvic Pain; Chronic Pain

ARMS (3):
- Mindfulness-based treatment (Experimental): The mindfulness-based psychological treatment consists of 10 weekly group sessions of 3 hours duration. The treatment is based on Mindfulness-based stress reduction (MBSR), Mindfulness-based cognitive therapy (MBCT) and Acceptance and commitment therapy (ACT). The intervention is partly manualized to accommodate demands of methodology, accuracy and repeatability. The group sessions will include:
  1. mindfulness-training (including meditation and yoga),
  2. therapy based on ACT, and
  3. patient-education in themes specifically targeted living with endometriosis-related chronic pelvic pain.
  Interventions: Other: Mindfulness-based psychological treatment
- Non-specific treatment (Experimental): The non-specific general psychological treatment is matched the mindfulness-based psychological treatment and consists of 10 weekly group sessions of 3 hours duration. The treatment is based on Client-centered therapy. The intervention is partly manualized to accommodate demands of methodology, accuracy and repeatability. The group sessions will include:
  1. relaxation and physical training,
  2. therapy based on the non-specific factors of psychological treatment which emphasize a focus on the relation and alliance between the therapist and the client and the therapist being a warm empathic, non-directive and unconditionally accepting support, and
  3. patient-education in themes specifically targeted living with endometriosis-related chronic pelvic pain.
  Interventions: Other: Non-specific psychological treatment
- Waiting list control (No Intervention): Participants in this arm will be on the waiting list to participate in one of the two experimental treatments after a period of six months. Participants will receive medical treatment as usual in this period.

INTERVENTIONS:
Other: Mindfulness-based psychological treatment
  Arms: Mindfulness-based treatment
Other: Non-specific psychological treatment
  Arms: Non-specific treatment

SUMMARY:
This study evaluates the effects of psychological treatment on pain, quality of life and work ability among women with endometriosis related chronic pelvic pain in a three-armed, randomised study. One group will receive mindfulness-based psychological treatment, the second group will receive a non-specific general psychological treatment (a psychological placebo) and the third group will be a waiting list control (treatment as usual).

ELIGIBILITY:
Inclusion Criteria:

* Endometriosis diagnosed by laparoscopy or MRI.
* Moderate to severe endometriosis-related chronic pelvic pain.
* Relevant clinical and surgical treatment according to the European Society of Human Reproduction and Embryology (ESHRE) guidelines for endometriosis have been tried.

Exclusion Criteria:

* Fibromyalgia, Colitis Chron or Colitis Ulcerosa
* Severe psychiatric diagnosis
* Pregnancy or planned pregnancy during the study period

Ages: 18 Years to 47 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2016-03; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Pelvic pain measured on Numeric Rating Scale | Change from pre-intervention to post-intervention (12 weeks)
  Pain intensity (sensory) and pain unpleasantness (affective) will be measured on Numeric Rating Scale (NRS: 0 = no pain till 10 = worst pain imaginable) in a daily pain diary.

SECONDARY OUTCOMES:
Quality of life measured by the Endometriosis Health Profile 30 questionnaire | Change from pre-intervention to post-intervention (12 weeks)
  Quality of life will be measured by the Endometriosis Health Profile 30 questionnaire (EHP-30) which is a patient generated questionnaire that measure endometriosis-related quality of life
Endometriosis related symptoms measured on Numeric Rating Scale | Change from pre-intervention to post-intervention (12 weeks)
  Dyspareunia, Dysmenorrhea, Dyschezia, Dysuria, Tiredness, Constipation, Diarrhea, Nausea and Vomiting will be measured on Numeric Rating Scale (NRS: 0 = no pain till 10 = worst pain imaginable) in a weekly diary.
Pain acceptance measured by Chronic Pain Acceptance Questionnaire | Change from pre-intervention to post-intervention (12 weeks)
  Pain acceptance measured by Chronic Pain Acceptance Questionnaire
Work Ability measured by the Work Ability Index | Change from pre-intervention to post-intervention (12 weeks)
  Work ability will be measured by the Work Ability Index (WAI) which is a questionnaire used to measure changes in work ability due to a specific intervention
Vaginal pressure pain detection threshold (PPDT) examined with a modified pressure algometer (palpometer) | Change from pre-intervention to post-intervention (12 weeks)
  Vaginal pressure pain detection threshold (PPDT) will be examined with a modified pressure algometer (palpometer) applicable for intravaginal pelvic floor muscle examination.

OTHER OUTCOMES:
Psychological flexibility measured by the Acceptance and Action Questionnaire-II | Change from pre-intervention to post-intervention (12 weeks)
  Psychological flexibility will be measured by the Acceptance and Action Questionnaire-II (AAQ-II)
Mindfulness measured by the Five Facet Mindfulness Questionnaire | Change from pre-intervention to post-intervention (12 weeks)
  Mindfulness will be measured by the Five Facet Mindfulness Questionnaire (FFMQ)

CONTACTS AND LOCATIONS:
Overall Officials: Axel Forman, Study Chair — Aarhus University Hospital; Lene Vase, Study Director — University of Aarhus; Karina E Hansen, Principal Investigator — University of Aarhus
Locations (3):
- Denmark (3):
  - Aarhus University Hospital, Department of Obstetrics and Gynecology, Aarhus N
  - Copenhagen University Hospital, Department of Gynaecology, Copenhagen
  - North Denmark Regional Hospital, Hjørring

REFERENCES:
- [Derived] Hansen KE, Brandsborg B, Kesmodel US, Forman A, Kold M, Pristed R, Donchulyesko O, Hartwell D, Vase L. Psychological interventions improve quality of life despite persistent pain in endometriosis: results of a 3-armed randomized controlled trial. Qual Life Res. 2023 Jun;32(6):1727-1744. doi: 10.1007/s11136-023-03346-9. Epub 2023 Feb 17. PMID 36797461